CLINICAL TRIAL: NCT01984320
Title: Combining Cabergoline and Coasting in Gonadotropin Releasing Hormone(GnRH)Agonist Protocol in Intracytoplasmic Sperm Injection (ICSI) to Prevent Ovarian Hyperstimulation Syndrome (OHSS): a Randomized Clinical Trial
Brief Title: Cabergoline and Coasting to Prevent OHSS
Acronym: OHSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Ahmed Bassiouny, MD, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 92013
Record Dates: First submitted 2013-10-31; First posted 2013-11-14 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: OHSS
Keywords: OHSS; ICSI; Coasting; Cabergoline
MeSH Terms: interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coasting (Active Comparator): In their ICSI cycle patients will continue their agonist treatment while stopping the human menopausal gonadotropin (hMG) injections for 1 to 3 days until drop of estradiol to a safe level to prevent OHSS. Early OHSS is assessed at day of embryo transfer and 7 days after this date. Late OHSS is assessed 14 days after embryo transfer.
  Interventions: Procedure: ICSI
- Cabergoline (Active Comparator): In their ICSI cycle patients will take 0.25 mg of cabergoline daily for 8 days from HCG triggering day to prevent OHSS. Early OHSS is assessed at day of embryo transfer and 7 days after this date. Late OHSS is assessed 14 days after embryo transfer.
  Interventions: Procedure: ICSI
- Coasting and Cabergoline (Active Comparator): In their ICSI cycle patients will continue their agonist treatment while stopping the human menopausal gonadotropin (hMG) injections for 1 day plus receiving 0.25 mg of cabergoline daily for 8 days from HCG triggering day to prevent OHSS. Early OHSS is assessed at day of embryo transfer and 7 days after this date. Late OHSS is assessed 14 days after embryo transfer.
  Interventions: Procedure: ICSI

INTERVENTIONS:
Procedure: ICSI — Long luteal GnRH agonist protocol: patients will receive GnRH agonist from day 21 of the previous cycle of stimulation and then on day 3 of the stimulation cycle they will start hMG injections with 225 IU/day. Folliculometry will start on day 6 stimulation by vaginal ultrasound. Estradiol levels will be measured on day 8, 10 and 12 of stimulation if appropriate. According to ultrasound and estradiol level patients will be randomized to either one of the study arms. When ready final triggering will be done by human chorionic gonadotropin (10000 IU) and oocyte collection is done at 36 hour from triggering. Embryo transfer is then done 3 days afterwards with ultrasound guidance.

SUMMARY:
The effectiveness of cabergoline to prevent moderate-severe OHSS to coasting.

DETAILED DESCRIPTION:
To randomly compare three study groups under a high risk of developing OHSS to one of three arms of management, either coasting for 1 to 3 days or receiving cabergoline for 8 days or coasting for 1 day plus receiving cabergoline for 8 days in ICSI patients following the long luteal GnRH agonist protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age <or= 35, BMI <or= 30
2. Long protocol GnRH agonist cycles
3. Estradiol level on day of HCG >or= 3500 pg/ml
4. Retrieving more than 15 oocytes

Exclusion Criteria:

1. Male factor
2. Uterine factor

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Rate and degree of OHSS (composite outcome) | 14 days
  Symptoms of nausea, vomiting, shortness of breath, abdominal pain,abdominal distension. Ovarian size and fluid in douglas pouch by ultrasound. Haematocrit, total leucocytic count, creatinine and Estradiol level as biochemical markers. Early OHSS first 9 days after ovum pickup and late is after 9 days till 14 days (time of pregnancy test)

SECONDARY OUTCOMES:
Number of oocytes | 1 day
  Number of oocytes collected on the day of oocyte collection

OTHER OUTCOMES:
Number of Metaphase II (MII) oocytes | 1 day
  Number of MII oocytes collected on the day of oocyte collection
Fertilization rate | 2 days
  Number of embryos that show signs of fertilization in each patient
Number of embryos | 3 to 5 days
  Number of embryos assessed for embryo transfer in each patient
Implantation rate | 5 weeks
  the ratio of the number of gestational sacs to the number of embryos transferred
Chemical pregnancy rate | 14 days
  The patients who have a positive quantitative Beta human chorionic gonadotrophin (BHCG) and do not continue their pregnancy with a drop in the result and start of menstruation
Clinical pregnancy rate | 28 days
  patients who show an intra-uterine gestational sac with positive fetal pulsations on ultrasound 14 days after their pregnancy test
Early miscarriage rate | 12 weeks
  pregnancy loss in the first 12 weeks of gestation
Ongoing pregnancy rate | 12 weeks
  pregnancies going beyond 12 weeks of gestation
Live birth rate | 40 weeks
  live births occuring

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Roushdy, MD, Study Chair — Cairo University
Locations (1):
- IVF centre, Obstetrics and Gynaecology Department, Cairo University Hospitals (Kasr EL Aini), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esinler I, Bozdag G, Karakocsokmensuer L. Preventing ovarian hyperstimulation syndrome: cabergoline versus coasting. Arch Gynecol Obstet. 2013 Nov;288(5):1159-63. doi: 10.1007/s00404-013-2875-z. Epub 2013 May 16. PMID 23677417
- [Derived] Bassiouny YA, Dakhly DMR, Bayoumi YA, Salaheldin NM, Gouda HM, Hassan AA. Randomized trial of combined cabergoline and coasting in preventing ovarian hyperstimulation syndrome during in vitro fertilization/intracytoplasmic sperm injection cycles. Int J Gynaecol Obstet. 2018 Feb;140(2):217-222. doi: 10.1002/ijgo.12360. Epub 2017 Nov 9. PMID 29055130